CLINICAL TRIAL: NCT05878522
Title: A Phase 1, Randomized, Double-blind, Sponsor-Open, Placebo- and Positive-Controlled Crossover Study to Investigate the Effect of Multiple Doses of Sisunatovir on QTc Interval in Healthy Adult Participants
Brief Title: A Study to Investigate the Effects of Sisunatovir on QTc Interval in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C5241015
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — sisunatovir; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Single Group, Crossover study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sisunatovir and placebo oral capsules will be prepared in the CRU by 2 operators, 1 of whom is an unblinded pharmacist. Sisunatovir and placebo will be administered in blinded fashion to the subject.
  Moxifloxacin 400 mg tablets will be packaged in an open-label manner at the CRU in the individual dosing containers by 2 operators, 1 of whom is an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, practitioner, or pharmacist).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): 6 capsules of sisunatovir administered Q12 hours for 5 doses
  Interventions: Drug: sisunatovir
- Treatment B (Placebo Comparator): 6 capsules of placebo administered Q12 hours for 5 doses
  Interventions: Drug: placebo
- Treatment C (Active Comparator): 6 capsules of placebo administered Q12 hours for 4 doses, followed by a single tablet of moxifloxacin
  Interventions: Drug: moxifloxacin
- Treatment D (Experimental): 7 capsules of sisunatovir administered Q12 hours for 5 doses
  Interventions: Drug: sisunatovir

INTERVENTIONS:
Drug: sisunatovir — 6 capsules administered Q12 hours for 5 doses
  Other Names: PF-07923568
  Arms: Treatment A
Drug: placebo — 6 capsules administered Q12 hours for 5 doses
  Arms: Treatment B
Drug: moxifloxacin — 6 capsules of placebo administered Q12 hours for 4 doses, followed by a single tablet of moxifloxacin
  Arms: Treatment C
Drug: sisunatovir — 7 capsules administered Q12 hours for 5 doses
  Other Names: PF-07923568
  Arms: Treatment D

SUMMARY:
The purpose of the study is to investigate the effects of multiple oral doses of sisunatovir on QTc Interval.

This study is seeking participants who:

* are male or female of 18 years of age or older
* are examined to be healthy All participants will receive Treatment A, B, and C in a randomized order based on 6 possible sequences. All treatments will be taken by mouth. Participants assigned to treatment A will receive 5 oral doses of sisunatovir administered Q12 hours over 3 days in a fed state. Participants assigned to treatment B will receive 5 oral doses of matching placebo administered Q12 hours over 3 days in a fed state. Participants assigned to treatment C will receive 4 oral doses of placebo administered Q12 hours for 2 days followed by a single dose of 400 mg moxifloxacin on the morning of Day 3.

All participants will remain in the study clinic for 4 days for each treatment, for safety review, laboratory collections, and to assess how the study medicine affects QTc intervals.

All participants selected in the study will be required to go through a screening period up to 28 days. A screening period is the time during which a few participants are examined to see whether they are fit for the study. During this period, the participant's medical history and past and current medications will be reviewed. A series of tests will also be performed to see if they are good to be selected for the study. If the participant meets all required criteria and are interested in continuing, the participant will be brought into the study clinic to stay overnight for 4 days for each treatment. On day 4, the participant will be discharged. About 28 to 35 days after discharge following the final treatment, the participant will be contacted for a follow up visit either in person or by telephone. This is to check up on how the participant is doing and to conclude the study.

ELIGIBILITY:
Inclusion Criteria: for healthy volunteers:

* Body Mass Index (BMI) of 17.5 to 32 kg/m2, inclusive, and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent.
* At screening, no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, including blood pressure (BP) and pulse rate measurement, standard 12-lead electrocardiogram (ECG) and clinical laboratory tests.

  --Exclusion criteria for all participants:
* Any condition or surgery possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection)
* Those with increased risk if dosed with moxifloxacin
* Self-reported history or risk factors for QT prolongation or torsades de pointes, congenital deafness, family history of cardiac arrest or suggest death, and family history of long QT syndrome
* Positive human immunodeficiency virus (HIV) antibodies
* Positive drug or alcohol test
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility-estimated glomerular filtration rate (GFR) <60 mL/min/1.73m2 at screening
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Participants with an average QTc interval >450 milliseconds (ms) will not be allowed to participate in the study. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* GFR <60 mL/min/1.73m2 based on CKD-EPI equation
* AST or ALT level ≥1.5 x upper limit normal (ULN)
* Gamma-GT> 1.2 x ULN
* Alkaline phosphatase > 1.2 x ULN
* Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at a single site in the United States. A total of 43 participants were assigned in this study.
Groups:
- Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo: Healthy participants administered 5 doses of sisunatovir 300 milligram (mg) capsule orally every 12 hours (Q12) over 3 days in a fed condition in Period 1. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 2. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg: Healthy participants administered 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in Period 1. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 2. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 3. There was washout period of minimum 7 days between doses.
- Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo: Healthy participants administered 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 1. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 2. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg: Healthy participants administered 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 1. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 2. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 3. There was washout period of minimum 7 days between doses.
- Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo: Healthy participants administered 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 1. Followed by 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in Period 2. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo: Healthy participants administered 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 1. Followed by 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 2. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg: Healthy participants administered 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 1. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 2. Followed by 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg: Healthy participants administered 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 1. Followed by 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 2. Followed by 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg: Healthy participants administered 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 1. Followed by 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in Period 2. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 3. There was washout period of minimum 7 days between doses.
- Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg: Healthy participants administered 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 1. Followed by 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 2. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 3. There was washout period of minimum 7 days between doses.
- Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg: Healthy participants administered 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 1. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 2. Followed by 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
- Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg: Healthy participants administered 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in Period 1. Followed by 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in Period 2. Followed by 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in Period 3. There was washout period of minimum 7 days between doses.
Period: Treatment Period- 1 (3 Days)
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg
Started | 2 | 2 | 5 | 5 | 2 | 4 | 2 | 5 | 3 | 5 | 3 | 5
Completed | 2 | 2 | 5 | 5 | 2 | 4 | 2 | 5 | 2 | 5 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — no longer meets eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period-1 (7 Days)
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg
Started | 2 | 2 | 5 | 5 | 2 | 4 | 2 | 5 | 2 | 5 | 3 | 5
Completed | 2 | 2 | 5 | 5 | 2 | 4 | 2 | 5 | 2 | 5 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period- 2 (3 Days)
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg
Started | 2 | 2 | 5 | 5 | 2 | 4 | 2 | 5 | 2 | 5 | 3 | 5
Completed | 1 | 1 | 5 | 4 | 1 | 4 | 2 | 5 | 2 | 4 | 3 | 5
Not Completed | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period-2 (7 Days)
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg
Started | 1 | 1 | 5 | 4 | 1 | 4 | 2 | 5 | 2 | 4 | 3 | 5
Completed | 1 | 1 | 5 | 4 | 1 | 4 | 2 | 5 | 2 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period- 3 (3 Days)
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg
Started | 1 | 1 | 5 | 4 | 1 | 4 | 2 | 5 | 2 | 4 | 3 | 5
Completed | 1 | 1 | 5 | 4 | 1 | 4 | 2 | 5 | 2 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sisunatovir 300 mg Followed by (=>) Placebo + Moxifloxacin 400mg => Placebo | Sisunatovir 300 mg => Placebo => Placebo + Moxifloxacin 400 mg | Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg => Placebo | Sisunatovir 350 mg => Placebo => Placebo + Moxifloxacin 400 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg | Placebo => Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg | Placebo => Sisunatovir 300 mg => Placebo + Moxifloxacin 400 mg | Placebo => Sisunatovir 350 mg => Placebo + Moxifloxacin 400 mg | Placebo + Moxifloxacin 400 mg => Sisunatovir 300 mg => Placebo | Placebo + Moxifloxacin 400 mg => Sisunatovir 350 mg => Placebo | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 300 mg | Placebo + Moxifloxacin 400 mg => Placebo => Sisunatovir 350 mg | Total
Number analyzed (Participants) | 2 | 2 | 5 | 5 | 3 | 5 | 3 | 5 | 2 | 4 | 2 | 5 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.00 (7.07) | 37.00 (7.07) | 42.20 (13.57) | 41.00 (10.79) | 48.67 (11.72) | 45.40 (11.72) | 50.00 (9.54) | 38.40 (14.43) | 37.00 (1.41) | 42.00 (11.28) | 60.00 (2.83) | 45.40 (16.09) | 43.30 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 15
  Male | 0 | 1 | 2 | 4 | 3 | 4 | 3 | 4 | 1 | 1 | 1 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 11
  Not Hispanic or Latino | 2 | 2 | 4 | 3 | 3 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 2 | 3 | 3 | 1 | 1 | 2 | 1 | 1 | 1 | 19
  White | 1 | 1 | 2 | 2 | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 4 | 18
  More than one race | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Placebo-Adjusted Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF) at Expected Maximum Concentration (Cmax) on Day 3 for Sisunatovir
Description: The relationship between sisunatovir plasma concentration and change from baseline in Fridericia's heart-rate corrected QT interval were analyzed using a model-based concentration-QTc analysis consistent with the Scientific White Paper on Concentration-QT Modeling. Baseline was defined as the mean of the 3 averages of the triplicate electrocardiogram (ECG) measurements taken before dosing on Day 1 within each period. Mean and CI statistics were based on the individual (within subject) corrected differences between sisunatovir and placebo exposures.
Time Frame: Baseline, Day 3
Population: The concentration QTc analysis set was defined as all participants randomized and treated with sisunatovir or placebo who had at least 1 pair of time-matched post-dose QT and sisunatovir plasma concentration values in at least 1 period of the study. For placebo treatment, the concentration was set to 0. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (90% Confidence Interval); unit: Milli seconds (msec)
Groups:
- Sisunatovir 300 mg: Healthy participants administered 5 doses of sisunatovir 300 mg capsule orally every Q12 over 3 days in a fed condition in any of the treatment periods.
- Sisunatovir 350 mg: Healthy participants administered 5 doses of sisunatovir 350 mg capsule orally every Q12 over 3 days in a fed condition in any of the treatment periods.
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg
Number analyzed (Participants) | 13 | 29
Milli seconds (msec) | 0.13 [-1.6 to 1.86] | -0.93 [-3.44 to 1.58]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An adverse event was considered a Treatment-Emergent Adverse Event (TEAE) if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time but before the end of the study were considered as TEAEs.
Time Frame: From start of treatment on Day 1 up to 38 days after last dose of study drug (maximum up to 10 weeks)
Population: Safety analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Healthy participants administered 5 doses of matching placebo orally administered every 12 hours for 2 days in a fed condition in any of the treatment periods.
- Placebo + Moxifloxacin 400 mg: Healthy participants administered 4 doses of matching placebo orally administered every Q12 hours for 2 days and a single dose of moxifloxacin 400 mg tablets administered orally on the morning of Day 3 in any of the treatment periods.
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg | Placebo | Placebo + Moxifloxacin 400 mg
Number analyzed (Participants) | 13 | 29 | 41 | 39
Participants | 8 | 9 | 10 | 12

3. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram Parameters
Description: Standard 12-lead ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, QTcF, and QRS complex. Clinical significance was determined based on investigator's discretion. Baseline of ECG parameters was defined as average of the triplicate ECGs collected at each time point before dosing on Day 1 within each period.
Time Frame: From Baseline up to Day 23
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg | Placebo | Placebo + Moxifloxacin 400 mg
Number analyzed (Participants) | 13 | 29 | 41 | 39
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Meeting Pre-defined Criteria for Vital Signs
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured with the participant in a supine position after at least 5 minutes of rest. Vital signs were categorized as 1) supine diastolic blood pressure (DBP) minimum (min) less than (<)50 and maximum (max) increase greater than or equal to (>=) 20 millimeter of mercury (mmHg); 2) supine systolic blood pressure (SBP) max. decrease >=20 and min. <90 (mmHg).
Time Frame: From Baseline up to Day 23
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg | Placebo | Placebo + Moxifloxacin 400 mg
Number analyzed (Participants) | 13 | 29 | 41 | 39
Participants
  Supine diastolic blood pressure (mmHg) min. <50 | 0 | 2 | 1 | 2
  Supine diastolic blood pressure (mmHg) max. increase >=20 | 1 | 0 | 0 | 0
  Supine systolic blood pressure (mmHg) max. decrease >=20 | 0 | 1 | 0 | 2
  Supine systolic blood pressure (mmHg) min. <90 | 0 | 0 | 2 | 2

5. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Abnormalities
Description: The clinical laboratory tests include hematology, chemistry, urinalysis and other tests. Following parameters were analyzed for laboratory assessments: Hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); Chemistry: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Albumin, Alkaline Phosphatase, Total Bilirubin, Creatinine, Uric Acid, Sodium, Potassium; Glucose(Fasting), Urea, Chloride, Bicarbonates, Total protein; Urinalysis: (decimal logarithm of reciprocal of hydrogen ion activity )[pH], Glucose, Protein, Blood, Ketones, Nitrites, Leukocyte esterase; Others tests: Pregnancy test, Urine drug screening, Covid-19 testing. Clinically significant laboratory abnormality findings were based on investigator discretion.
Time Frame: From Baseline up to Day 23
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg | Placebo | Placebo + Moxifloxacin 400 mg
Number analyzed (Participants) | 13 | 29 | 40 | 39
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in QTcF of Moxifloxacin and Placebo at 3, 4 and 5 Hours Post-Dose of Day 3
Description: Change from baseline in QTcF intervals were analyzed using a MMRM model with sequence, period, treatment, time (post-dose timepoint) and treatment by time interaction as fixed effect, participants within sequence as a random effect and baseline QTcF as a covariate. A compound symmetry covariance matrix was fitted to the repeated times within participant and the Kenward-Roger approximation was used for estimating degrees of freedom.
Time Frame: Baseline, 3, 4 and 5 hours post-dose on Day 3
Population: ECG analysis set included all participants who were randomized and treated who have at least 1 post-dose ECG measurement in at least 1 period. This was planned to be reported in moxifloxacin and placebo as pre-specified in protocol. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- PLACEBO + MOXIFLOXACIN 400 MG TABLET: Healthy participants were administered oral dose of placebo with a single oral dose of Moxifloxacin 400 mg tablet in any of the treatment periods.
Arm/Group | PLACEBO + MOXIFLOXACIN 400 MG TABLET | Placebo
Number analyzed (Participants) | 39 | 40
msec
  3 hours post-dose | 3.97 [1.88 to 6.05] | -7.77 [-9.86 to -5.68]
  4 hours post-dose | 6.63 [4.54 to 8.72] | -4.72 [-6.81 to -2.63]
  5 hours post-dose | 6.84 [4.75 to 8.93] | -1.52 [-3.61 to 0.57]
Statistical Analysis 1: Comparison: PLACEBO + MOXIFLOXACIN 400 MG TABLET; 3- hours post-dose; Test type: Other; LS Mean difference = 11.73, 90% CI 2-sided [8.89 to 14.58]
Statistical Analysis 2: Comparison: PLACEBO + MOXIFLOXACIN 400 MG TABLET; 4-hours post-dose; Test type: Other; LS Mean difference = 11.35, 90% CI 2-sided [8.50 to 14.20]
Statistical Analysis 3: Comparison: PLACEBO + MOXIFLOXACIN 400 MG TABLET; 5-hours post-dose; Test type: Other; LS Mean difference = 8.35, 90% CI [5.51 to 11.20]

ADVERSE EVENTS:
Time Frame: From start of treatment on Day 1 up to 38 days after last dose of study drug (maximum up to 10 weeks)
Description: Safety population included all participants randomly assigned and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Arm/Group | Sisunatovir 300 mg | Sisunatovir 350 mg | Placebo | Placebo + Moxifloxacin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/29 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/29 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 8/13 | 8/29 | 4/41 | 7/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sisunatovir 300 mg (N=13) | Sisunatovir 350 mg (N=29) | Placebo (N=41) | Placebo + Moxifloxacin 400 mg (N=39)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Brain fog (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT05878522/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT05878522/SAP_001.pdf